CLINICAL TRIAL: NCT06989398
Title: Cluster RCT of the WHO's Advancing Supervisor Capabilities for Mental Health at Work (ASCEND) in Dutch Small and Medium-sized Enterprises (SMEs)
Brief Title: Implementation of the ASCEND Training for Supervisors in Dutch Small and Medium-sized Enterprises (SMEs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: World Health Organization (Other); University of Copenhagen (Other); University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Mark van Vugt, Full Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024.0846; ADVANCE (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2025-05-06; First posted 2025-05-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: Occupational Health; Stress; Burnout; Mental Health Conditions; Sickness Absence
Keywords: Workplace mental health; Occupational stress; Sickness absence; Supervisors; Line managers; Absenteeism; Presenteeism; Employee well-being; Workplace intervention; Manager training; ASCEND; Advancing Supervisors' Capacity for Mental Health at Work
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Intervention Model Description: The trial has cluster-randomized study design, meaning that the organizations (i.e., SMEs) that take part in the study will form clusters that will be randomized into either the intervention or control group. This way every participating employee from a SME is part of the same group.
  The SMEs will be randomized using limited block size that varies randomly (i.e., 4, 6, or 8 SMEs per block) across (1) ASCEND (n=37) or (2) Waitlist (n=37), with an equal probability of assignment to each group (allocation ratio 1:1).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advancing Supervisors' Capacity for Mental Health at Work (ASCEND) (Experimental): The intervention will consist of a training that incorporates evidence-based content and interactive exercises. Advancing Supervisors' Capacity for Mental Health at Work (ASCEND) covers five core topics designed to equip supervisors with the knowledge and practical skills needed to effectively support the mental health of their employees. The full training is delivered over approximately 8 hours in an in-person group setting. Trainings are facilitated by a trained professional.
  Interventions: Behavioral: Advancing Supervisors' Capacity for Mental Health at Work (ASCEND)
- Waitlist (No Intervention): Supervisors from organizations in the waitlist arm will receive no training during the trial. They will be provided with the ASCEND training approx. 6 months after baseline, after the last follow-up.

INTERVENTIONS:
Behavioral: Advancing Supervisors' Capacity for Mental Health at Work (ASCEND) — The intervention will consist of a training that incorporates evidence-based content and interactive exercises. Advancing Supervisors' Capacity for Mental Health at Work (ASCEND) covers five core topics designed to equip supervisors with the knowledge and practical skills needed to effectively support the mental health of their employees. The full training is delivered over approximately 8 hours in an in-person group setting. Trainings are facilitated by a trained professional.
  To support learning and skill application, participants will also receive a Manager Reference Booklet during the training. This booklet consolidates key information from the ASCEND training, serving both as a learning aid during the sessions and a practical, quick-reference tool afterward. It includes summaries of key concepts, tips, and exercises, along with space for participants to record notes.
  Other Names: Toolkit Mental Health for Supervisors; Toolkit Mentale Gezondheid voor Leidinggevenden
  Arms: Advancing Supervisors' Capacity for Mental Health at Work (ASCEND)

SUMMARY:
This cluster randomized controlled trial (cRCT) aims to evaluate the effectiveness of an in-person group intervention for workplace supervisors - Advancing Supervisors' Capacity for Mental Health at Work (ASCEND) - in Dutch Small and Medium-sized Enterprises (SMEs). The ASCEND intervention is designed to equip supervisors with the skills to: i) know when to support their workers; ii) how to direct workers to support, and iii) advocate for action on mental health at work.

The primary objectives of this project are to:

* Assess to what extent the novel, WHO-developed ASCEND intervention is effective in enhancing supervisors' confidence, responsiveness, mental health literacy, and SelfCare practices, and in reducing supervisor stigma towards mental health conditions within Dutch SMEs.
* Evaluate the impact of the ASCEND intervention on employee outcomes, including mental health and work-related outcomes among supervisees (i.e., subordinates), as well as overall organizational absenteeism rates.
* Identify barriers, facilitators, and key implementation and adoption indicators to support future opportunities for scaling up the ASCEND intervention in the context of Dutch SMEs.

Researchers will compare two groups to evaluate the effectiveness of the ASCEND intervention. One group will receive the training (the intervention group), while the other group will receive the training after the final follow-up period (the control group).

Data will be collected from both supervisors and their supervisees (i.e., subordinates) via online questionnaires at various time points. In addition, general organizational information, including absenteeism rates, will be gathered through a representative from each participating organization.

To further explore the feasibility of scaling up the ASCEND intervention within the Netherlands, qualitative data will be collected through interviews and/or focus group discussions.

DETAILED DESCRIPTION:
Small and Medium-sized enterprises (SMEs) often lack the resources to effectively address the negative consequences of work-related stressors (e.g., high workplace digitalization). Moreover, supervisors play a pivotal role in protecting employee well-being, yet they frequently report feeling poorly equipped to recognize and support employees experiencing mental health problems.

This project aims to evaluate the effectiveness of Advancing Supervisors' Capacity for Mental Health at Work (ASCEND), an in-person group intervention developed by the World Health Organization (WHO). The ASCEND intervention is designed to equip supervisors with the skills to: i) know when to support their workers; ii) how to direct workers to support, and iii) advocate for action on mental health at work.

The first phase of this study concerns a cluster randomized controlled trial (cRCT) comparing ASCEND and waitlist, where supervisors in the control group receive the intervention approx. 6 months after baseline. The second phase consists in the qualitative process evaluation that pertains individual interviews and/or focus group discussions.

In the first study phase, data will be collected through online questionnaires administered to supervisors and their supervisees (i.e., subordinates). Additionally, general organizational information, including absenteeism rates, will be gathered from a designated representative within each organization. Supervisors in the intervention group will complete surveys at baseline, immediately post-intervention, and at 1-month and 3-month follow-ups. Supervisors in the control group, as well as supervisees, will complete surveys at baseline, 1-month follow-up, and 3-month follow-up.

The primary outcome is supervisor confidence in supporting employees with mental health conditions at the 1-month follow-up. Secondary outcomes include supervisor responsiveness, stigma toward mental health conditions, mental health literacy, and SelfCare practices. Supervisees will be invited to provide exploratory outcome data on perceived supervisor responsiveness, perceived StaffCare, psychological distress, help-seeking intentions, work stress, absenteeism, and presenteeism. Additionally, general absenteeism figures for the participating SMEs will be collected.

The study aims to recruit 74 SMEs, randomly allocated to either the ASCEND intervention group (n = 37) or the waitlist control group (n = 37). Each SME is expected to enrol at least two supervisors, resulting in a total sample of 148 managers for this study phase. Sample size calculations indicate that a minimum of 60 SMEs is required to detect a significant increase in supervisor confidence at 1-month follow-up with an effect size of Cohen's d = 0.59, accounting for 20% attrition (power = 0.80, two-sided alpha = 0.05, ICC = 0.01).

In the second study phase, a process evaluation will be conducted to assess factors such as intervention acceptability, appropriateness, barriers, and facilitators to implementation. Qualitative data will be gathered through post-intervention online surveys and interviews with a sample of supervisors, as well as relevant other stakeholders.

This study is part of the larger EU H2022-ADVANCE project, which aims to improve the mental health of vulnerable populations in Europe.

ELIGIBILITY:
Inclusion for SMEs:

* Having 10 to 250 employees
* Being located in the Netherlands

In case of insufficient recruitment among SMEs, a mitigation strategy is to recruit individual departments from larger organizations.

Eligibility criteria for individual participants:

Supervisors are included if they fit the following inclusion criteria:

* 18 years or older
* Working in an organization in the Netherlands
* Sufficient mastery (written and spoken) of the language in which the ASCEND intervention is being delivered (i.e., Dutch or English)
* Written informed consent before entering the study
* Supervise at least 1 supervisee within the same organization

Supervisees are included if they fit the following inclusion criteria:

* 18 years or older
* Have a direct supervisor who is participating in ASCEND (either intervention or control group)
* Sufficient mastery of English or Dutch
* Written informed consent before entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Supervisor confidence in supporting employees with mental health conditions | Change from baseline to 1-hour post-intervention, 1 month, and 3 months
  Confidence in supporting employees with mental health conditions will be measured among supervisors using a 6-item scale used in other trials that investigated a similar intervention. Participants will be asked to rate their degree of confidence from 1 (not confident at all) to 5 (extremely confident) for various activities that are related to the construct of supporting employee mental health. A mean score will be calculated by averaging participants' ratings across all items. Scores range from 1 to 5, with a higher score indicating more confidence.

SECONDARY OUTCOMES:
Supervisor responsiveness to employee mental health conditions | Change from baseline to 1 month and 3 months
  Responsiveness to mental health conditions will be measured among supervisors using a 6-item scale used in earlier trials investigating a similar intervention. Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. A mean score will be calculated by averaging participants' ratings across all items. Scores range from 1 to 5, with a higher score indicating a better responsiveness.
Supervisor stigma towards mental health conditions | Change from baseline to 1-hour post-intervention, 1 month, and 3 months
  Stigma towards mental health conditions will be measured among supervisors using the 12-item Stigma Toward Employee Depression Scale. Items are adjusted to fit a broader range of mental health conditions, instead of depression only. Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. A mean score will be calculated by averaging participants' ratings across all items. Scores range from 1 to 5, with a higher score indicating more stigma.
Supervisor SelfCare | Change from baseline to 1 month and 3 months
  SelfCare will be measured among supervisors using a construct originating from the Health-oriented Leadership framework. The full SelfCare scale consists of 3 subscales (i.e., awareness, values, and behavior), but this trial focuses only on the behaviors. From the behavior items, 3 items are chosen. Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. A mean score will be calculated by averaging participants' ratings across all items. Scores range from 1 to 5, with a higher score indicating better SelfCare.
Supervisor mental health literacy | Change from baseline to 1-hour post-intervention and 1 month
  Mental health literacy will be measured among supervisors using vignette-based questions, based on vignettes from the Mental Health Literacy (MHL) scale. Supervisors will respond to open-ended questions about how they would handle each of the workplace scenarios described in the vignettes. Responses will be scored at a later stage. Each vignette-question will receive a score from 0 to 2, with higher scores reflecting higher mental health literacy.
Implementation indicator: acceptability | 1-hour post-intervention
  The implementation indicator of acceptability is measured post-intervention through self-reported item(s). Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. Higher scores indicate higher acceptability.
Implementation indicator: appropriateness | 1-hour post-intervention
  The implementation indicator of appropriateness is measured post-intervention through self-reported item(s). Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. Higher scores indicate higher appropriateness.

OTHER OUTCOMES:
Perceived supervisor responsiveness to mental health conditions | Change from baseline to 1 month and 3 months
  Perceived supervisor responsiveness to mental health conditions will be measured among supervisees, using the same construct (i.e., 'Supervisor responsiveness to mental health conditions') that is measured among supervisors. Two items of the original will be included and adjusted to fit the context of the supervises. Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. A mean score will be calculated by averaging participants' ratings across all items. Scores range from 1 to 5, with a higher score indicating a higher perceived responsiveness.
Perceived StaffCare | Change from baseline to 1 month and 3 months
  StaffCare will be measured among supervisees using a construct originating from the Health-oriented Leadership framework. The full SelfCare scale consists of 3 subscales (i.e., awareness, values, and behavior), this trial focuses only on the behaviors. From the behavior items, some items are chosen to be included. Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. A mean score will be calculated by averaging participants' ratings across all items. Scores range from 1 to 5, with a higher score indicating better perceived StaffCare.
Supervisee psychological distress | Change from baseline to 1 month and 3 months
  Psychological distress will be measured among supervisees using the 6-item Kessler Psychological Distress Scale (K6). The K6 consists of 6 items asking people to rate their emotional states on a 5-point Likert scale ranging from 1 (none of the time') to 5 (all the time). Scores are summed and scores range from 0 to 24. Higher scores indicate increased non-specified psychological distress.
Supervisee help-seeking intentions | Change from baseline to 1 month and 3 months
  Help-seeking intentions will be measured among supervisees using the General Help Seeking Questionnaire. Participants are asked how likely it would be that they would seek help from 5 resources (e.g., direct supervisor, company mental health resources, doctor/GP, mental health professional, or other) on a scale ranging from 1 (very unlikely) to 5 (very likely), with higher scores indicating a greater intention to seek help.
Supervisee work stress | Change from baseline to 1 month and 3 months
  Work stress will be measured among supervisees using the 4-item job stress scale. Participants rate each item on a 5-point Likert scale with 1 (strongly disagree) to 5 (strongly agree) to what extent they agree with the statement. A mean score will be calculated by averaging participants' ratings across all items. Scores range from 1 to 5, with a higher score indicating higher levels of work-related stress.
Supervisee presenteeism | Change from baseline to 1 month and 3 months
  Presenteeism will be measured among supervisees using 1 item. Participants report the number of days they have been less productive than usual due to illness in the last 4 days in a text box. Higher scores indicate more unproductive days.
Supervisee absenteeism | Change from baseline to 1 month and 3 months
  Absenteeism will be measured among supervisees using 1 item. Participants answer this question by mentioning the number of days they have been absent due to illness in the last 4 weeks in a text box. Higher scores indicate more sick days.
General absenteeism | Change from 6 months before to 6 months after the trial's start
  General absenteeism rates will be recorded for the 6 months before and after the start of the trial. This will be reported by a representative of the organization.

CONTACTS AND LOCATIONS:
Overall Officials: Mark van Vugt, PhD, Principal Investigator — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: ADVANCE project website — https://advancementalhealth.ku.dk/